CLINICAL TRIAL: NCT02362061
Title: Thickness of the Junctional Zone Measured by 3D Ultrasound and Its Relation to the Success/Failure Implantation Rates in Assisted Reproduction Techniques
Brief Title: 3D Ultrasound Measurement of Junctional Zone Thickness and Its Relation to Implantation Success
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 128
Record Dates: First submitted 2015-02-07; First posted 2015-02-12 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Infertility
Keywords: junctional zone; implantation; three D ultraosund; Assisted Reproductive Technology; Pregnancy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pregnant: These patients are then assigned to receive fertility treatment (ovulation induction, ICSI, intrauterine insemination and IVF). They undergo a 3D vaginal ultrasound before treatment to measure the junctional zone thickness and followed up after treatment to determine the rate of implantation and they became pregnant
  Interventions: Radiation: 3D ultrasound
- Non pregnant: These patients are then assigned to receive fertility treatment (ovulation induction, ICSI, intrauterine insemination and IVF). They undergo a 3D vaginal ultrasound before treatment to measure the junctional zone thickness and followed up after treatment to determine the rate of implantation and they remained non pregnant
  Interventions: Radiation: 3D ultrasound

INTERVENTIONS:
Radiation: 3D ultrasound — ultrasound to measure the thickness of the junctional zone at day 21 of the cycle

SUMMARY:
100 patients aged 21-40 years old, diagnosed as primary or secondary infertility . These patients are then assigned to receive fertility treatment (ovulation induction, ICSI, intrauterine insemination and IVF). They undergo a 3D vaginal ultrasound before treatment to measure the junctional zone thickness and followed up after treatment to determine the rate of implantation.

ELIGIBILITY:
Inclusion Criteria:

* infertile women

Exclusion Criteria:

* congenital uterine anomalies medical disease contraindicating pregnancy

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 patients aged 21-40 years old, diagnosed as primary or secondary infertility due to the following causes of infertility; ( Pelvic Inflammatory disease, dysovulation , tubal infertility, unexplained infertility, combined infertility or due to male factor ).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 14 days after evaluation

SECONDARY OUTCOMES:
healthy pregnancy | 6 weeks after pregnancy confirmation by pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt